CLINICAL TRIAL: NCT05790291
Title: The Effect Of The Check List Developed For Drug Administration From Enteral Nutrition Tube On Administration Errors
Brief Title: Drug Administration From Enteral Nutrition Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emel Külekçi (Other)
Responsible Party: Sponsor-Investigator, Emel Külekçi, Lecturer, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021/29
Record Dates: First submitted 2023-02-16; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Intensive Care
Keywords: Enteral Tube; Enteral Drug Administration; Nurse; Medication Errors; Checklist
MeSH Terms: interventions — Checklist

STUDY DESIGN:
Intervention Model Description: randomized control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: First, the participants were blinded. Participants were randomized after the pretest and divided into two groups. No explanation was given to the participants about how many groups there were and which group they belonged to.
  Second, the observer was blinded. Video recording was taken by the researcher during the administration in calculating the error rates.
  The video recordings were watched one by one by an assistant researcher who did not know the groups, and the administration steps were marked on the observation form as true/false.
  Third, the statistician was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- checklist (Experimental): checklist
  Interventions: Other: Checklist
- no intervention (No Intervention): no intervention

INTERVENTIONS:
Other: Checklist — the experimental group will practice using the checklist
  Arms: checklist

SUMMARY:
Enteral nutrition protocols are applied in patients who do not have gastrointestinal dysfunction but in whom oral feeding is contraindicated. In these patients, where drug use is also necessary but alternative drug administration routes are not possible, drugs can be given to the patient through enteral nutrition tubes. However, there are studies reporting errors and complications during drug administration from the enteral nutrition tube. With the planned thesis study, it is aimed to develop an evidence-based checklist and to reduce the rate of errors and complications in drug administration through enteral feeding tube with this checklist.

DETAILED DESCRIPTION:
Enteral nutrition protocols are applied in patients who do not have gastrointestinal dysfunction but in whom oral feeding is contraindicated. In these patients, where drug use is also necessary but alternative drug administration routes are not possible, drugs can be given to the patient through enteral nutrition tubes.

When adding drugs to parenteral nutrition admixtures or using concomitant drugs from the same catheter, it has become a general rule to check for drug incompatibility. The same level of care is not taken in drug administration from the enteral nutrition tube. There are studies reporting errors and complications in enteral drug administration in the literature Today, one of the most important parts of corporate culture in healthcare is patient safety. Patient safety is all of the measures taken by health institutions and employees in these institutions in order to prevent the harm that health care services may cause to individuals. The main goal here is; It is the establishment of a system that will protect the patient from possible harm and eliminate the possibility of error due to errors that will prevent the occurrence of errors during care delivery.

The checklists used in recent years are also an evidence-based practice list and have become one of the effective methods used to prevent errors and reduce complications. A checklist standardizes the process, streamlines maintenance delivery, and improves performance to ensure all actions are covered. The checklist allows cross-checking what was done and in what order. These reassurances are important in situations where time is short and distractions.

With this study, it is aimed to develop an evidence-based checklist and to reduce the rate of errors and complications in drug administration through enteral feeding tube with this checklist.

ELIGIBILITY:
Inclusion Criteria:

* Being an intensive care nurse
* Have experience in administering enteral medication
* Administering enteral medication to an adult patient
* Agree to participate in the research

Exclusion Criteria:

* Administering enteral medication to a patient with fluid restriction
* Change of position
* Wanting to leave research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change in enteral drug administration error rates of nurses with an interval of 2 months | baseline and month 2
  First, the error rates of 69 nurses during enteral drug administration were calculated.
  Enteral medication was administered for approximately one month with the next intervention group (n=34) checklist. Finally, the error rates of 69 nurses during enteral drug administration were recalculated.
  Error rates were determined with a 19-item observation formula. Name of the form; Medication from Enteral Feeding Tube Observation Form for Applications The lowest error rate is 0%, the highest error rate is 100%.

SECONDARY OUTCOMES:
Change in enteral drug administration knowledge of nurses with an interval of 2 months | baseline and month 2
  First, the knowledge levels of 69 nurses on enteral drug administration were calculated.
  Then the intervention group (n=34) administered enteral medication for approximately one month along with the checklist. Finally, the knowledge levels of 69 nurses on enteral drug administration were recalculated.
  Knowledge levels were determined with a 20-item information form. Name of the form; It is an Information Evaluation Form for Drug Administrations from Enteral Feeding Tube.
  The lowest score is 0, the highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL KÜLEKCİ, Principal Investigator — PhD student
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demirkan K, Ekincioğlu AB. Enteral Beslenme Tüpünden İlaç Uygulanmasında İlaç Dozaj Şekillerinin Önemi. Journal of the Turkish Society of Intensive Care/Türk Yogun Bakim Dernegi Dergisi. 2016;14(1):1-8.
- [Background] Ekincioglu AB, Demirkan K. Clinical nutrition and drug interactions. Ulus Cerrahi Derg. 2013 Nov 14;29(4):177-86. doi: 10.5152/UCD.2013.112013. eCollection 2013. PMID 25931873
- [Background] Abu Hdaib N, Albsoul-Younes A, Wazaify M. Oral medications administration through enteral feeding tube: Clinical pharmacist-led educational intervention to improve knowledge of Intensive care units' nurses at Jordan University Hospital. Saudi Pharm J. 2021 Feb;29(2):134-142. doi: 10.1016/j.jsps.2020.12.015. Epub 2021 Jan 7. PMID 33679176
- [Background] Sari D, Kadifeli D, Akbiyik A, Taskiran N. Intensive care unit nurses' knowledge of medication administration via enteral tubes. Nurs Crit Care. 2018 May;23(3):141-146. doi: 10.1111/nicc.12335. Epub 2018 Feb 8. PMID 29424127
- [Background] Çelik S, Demiray Y, Tuğrul A, Köymen H, Coşkun Y, Doğru Ö, et al. Yoğun bakım hemşirelerinin enteral tüp aracılığıyla ilaç uygulamalarının değerlendirilmesi. Çağdaş Tıp Dergisi. 2014;4(1):18-25.
- [Background] Emami S, Hamishehkar H, Mahmoodpoor A, Mashayekhi S, Asgharian P. Errors of oral medication administration in a patient with enteral feeding tube. J Res Pharm Pract. 2012 Jul;1(1):37-40. doi: 10.4103/2279-042X.99677. PMID 24991587
- [Background] Özkan D, Yavuz Van Giersbergen M. Güvenli Cerrahi Kontrol Listesi Konusunda Ameliyathane Ekibinin Düşüncelerinin İncelenmesi. Turkiye Klinikleri J Surg Nurs-Special Topics Türkiye Klinikleri Cerrahi Hastalıkları Hemşireliği-Güvenli Cerrahi Uygulamaları Özel Sayısı. 2016;2(3):22-8
- [Background] Winters BD, Gurses AP, Lehmann H, Sexton JB, Rampersad CJ, Pronovost PJ. Clinical review: checklists - translating evidence into practice. Crit Care. 2009;13(6):210. doi: 10.1186/cc7792. Epub 2009 Dec 31. PMID 20064195
- [Background] Bankhead R, Boullata J, Brantley S, Corkins M, Guenter P, Krenitsky J, Lyman B, Metheny NA, Mueller C, Robbins S, Wessel J; A.S.P.E.N. Board of Directors. Enteral nutrition practice recommendations. JPEN J Parenter Enteral Nutr. 2009 Mar-Apr;33(2):122-67. doi: 10.1177/0148607108330314. Epub 2009 Jan 26. No abstract available. PMID 19171692
- [Background] Boullata JI, Carrera AL, Harvey L, Escuro AA, Hudson L, Mays A, McGinnis C, Wessel JJ, Bajpai S, Beebe ML, Kinn TJ, Klang MG, Lord L, Martin K, Pompeii-Wolfe C, Sullivan J, Wood A, Malone A, Guenter P; ASPEN Safe Practices for Enteral Nutrition Therapy Task Force, American Society for Parenteral and Enteral Nutrition. ASPEN Safe Practices for Enteral Nutrition Therapy [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jan;41(1):15-103. doi: 10.1177/0148607116673053. Epub 2016 Nov 5. PMID 27815525
- [Background] Bischoff SC, Austin P, Boeykens K, Chourdakis M, Cuerda C, Jonkers-Schuitema C, Lichota M, Nyulasi I, Schneider SM, Stanga Z, Pironi L. ESPEN guideline on home enteral nutrition. Clin Nutr. 2020 Jan;39(1):5-22. doi: 10.1016/j.clnu.2019.04.022. Epub 2019 May 30. PMID 31255350

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05790291/SAP_000.pdf
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT05790291/ICF_001.pdf